CLINICAL TRIAL: NCT04670081
Title: A Phase II Randomized, Double-blind, Active Placebo-controlled Parallel Group Trial to Examine the Efficacy and Safety of Psilocybin in Treatment-resistant Major Depression
Brief Title: Efficacy and Safety of Psilocybin in Treatment-Resistant Major Depression
Acronym: EPIsoDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Charite University, Berlin, Germany (Other); MIND Foundation gGmbH (Unknown); German Federal Ministry of Education and Research (Other Government); Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPIsoDE_01
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Treatment-resistant Depression
Keywords: Psilocybin; Major depressive disorder; MDD; Psychedelics; 5-HT2A; double-blind
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Psilocybin; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nicotinamide (Placebo Comparator): 1st dose: 100 mg Nicotinamide (Vitamin B3) - 2nd dose (after 6 weeks/after assessment of the primary endpoint): 25 mg Psilocybin
  Interventions: Drug: Psilocybin; Drug: Nicotinamide
- Psilocybin (low-dose) (Experimental): 1st dose: 5 mg Psilocybin - 2nd dose (after 6 weeks/after assessment of the primary endpoint): 25 mg Psilocybin
  Interventions: Drug: Psilocybin
- Psilocybin (high-dose) (Experimental): 1. 1st dose: 25 mg Psilocybin - 2nd dose (after 6 weeks/after assessment of the primary endpoint): 5 mg Psilocybin
  2. 1st dose: 25 mg Psilocybin - 2nd dose (after 6 weeks/after assessment of the primary endpoint): 25 mg Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 25 mg, p.o.
Drug: Psilocybin — 5 mg, p.o.
  Arms: Psilocybin (high-dose); Psilocybin (low-dose)
Drug: Nicotinamide — 100 mg, p.o.
  Arms: Nicotinamide

SUMMARY:
The study aims to investigate the safety and efficacy of oral psilocybin administered under supportive conditions in treatment-resistant major depression (TRD).

The study is a bi-centric, prospective, randomized, active placebo-controlled study investigating the effects of 25 mg and 5 mg (p.o.) psilocybin versus placebo (100 mg nicotinamide) in a psychotherapeutic context in 144 patients with TRD from moderate to severe degree (ICD-10 F32/F33). After giving written informed consent and down-titration of their monoaminergic medication under supervision of the treating psychiatrist and the study team, patients will be randomly assigned to one of four trial arms using an online randomization tool: 1) receiving placebo (100 mg nicotinamide) at the first session and the full dose (25 mg) at the second; 2) receiving the presumably sub-effective dose (5 mg) at the first session and the full dose (25 mg) at the second; 3a) receiving the full dose (25 mg) at the first session and 5 mg at the second; 3b) receiving the full dose at both sessions. The two dosing sessions are accompanied by three preparatory and four integration sessions.

Drug administration must occur under psychotherapeutic conditions. Two trained therapists (one male, one female) will be assigned to each patient and be present during each dosing, preparatory and integration sessions. We will follow the safety guidelines provided by Johnson et al. (2), including a thorough preparation, establishment of trust/rapport, a safe and pleasing physical environment and sufficient interpersonal support. For safety reasons and close monitoring, patients will stay hospitalized for one night after each dosing session (i.e. in-patient setting).

ELIGIBILITY:
Inclusion Criteria:

1. 25 to 65 years of age
2. Diagnosis of major depressive disorder (single and recurrent episodes) of moderate to severe degree (HAM-D score ≥ 17) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) without psychotic features. Included ICD-10 diagnoses are ICD-10: F32.1, F32.2, F33.1, F33.2.

   a. If single episode, duration must be ≥ 3 months.
3. Patients must meet criteria for treatment-resistance, defined as

   a. no adequate improvement despite two adequate courses of antidepressant treatment (6 weeks each, minimum) with drugs of different pharmacological classes in the current depressive episode. Augmentation with an add-on treatment counts as a second treatment.
4. Patients have discontinued any monoaminergic psychiatric medication (i.e. SRIs, antipsychotic medication) for at least 2 weeks before the first dosing session.

   1. Patients who are still on any monoaminergic psychiatric medication at screening must agree to down-titrate over an individualized down-titration schedule (minimum 2 weeks; if they have been taken Fluoxetine the down-titration phase should be minimum 5 weeks) in close supervision by their out-patient psychiatrist and the study team. The treating psychiatrist must agree to supervise and monitor the down-titration and to collaborate with the study team by signing a "treatment agreement form".
   2. If the treating psychiatrist refuses to monitor the down-titration, the patient has to agree to down-titrate under supervision of clinicians in the outpatient clinics of the two study sites or trial physicians and to come in for weekly monitoring visits.
5. The subjects are abstinent from alcohol (breathalyzer blood alcohol concentration (BAC) level 0.00) and a negative urine drug screen at days of dosing
6. The subject must be medically stable based on clinical laboratory tests, medical history, vital signs, and 12-lead ECG performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase. In 12-lead ECG, QTcF should be ≤ 450 ms for males or ≤ 470 ms for females and PR-interval < 220 ms at screening. A retest of an abnormal ECG value will be allowed once in the screening phase. Blood pressure will be the average of 2 measurements. The subject may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the subject's source documents and initialed by the investigator.
7. The subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
8. The subject must sign an informed consent form indicating that he/she understands the purpose of and procedures required for the study including peripheral biomarker monitoring (i.e. blood) and is willing to participate in the study.

Exclusion Criteria:

1. Currently comorbid or previously diagnosed DSM-5 diagnosis of a

   1. major depressive episode with psychotic features/major depressive disorder with psychotic features (ICD-10: F32.3)
   2. schizophrenia spectrum and other psychotic disorders, including schizotypal (personality) disorders, delusional disorder, brief psychotic disorder, schizophreniform disorder, schizoaffective disorder, substance/medication-induced psychotic disorder and psychotic disorder due to another medical condition (ICD-10: F20 - F29)
   3. bipolar and related disorders (ICD-10: F30/F31)
   4. cluster A personality disorders (paranoid personality disorder, schizoid personality disorder, schizotypal personality disorder) and/or borderline personality disorder (Patients will be carefully screened for presence of those personality disorders by using the SCID-5-PD)
   5. Post-traumatic stress disorder (PTSD; ICD-10: F43.1)
2. A family history (first-degree relative) of psychosis and/or bipolar disorder
3. The subject has a current or recent history of clinically significant suicidal ideation within the past 6 months, corresponding to a score of 4 (active suicidal ideation with some intent to act, without specific plan) or 5 (active suicidal ideation with specific plan and intent) for ideation on the C-SSRS, or a history of suicidal behavior within the past 1 year, as validated by the C-SSRS at screening. Subjects with a prior suicide attempt of any sort, or prior serious suicidal ideation/plan > 6 months ago, should be carefully screened for current suicidal ideation and only included at the discretion of the investigator.
4. Current comorbid psychiatric diagnosis except their major diagnosis (inclusion criterion 3) in form of

   a. Diagnoses mentioned under exclusion criterion 1) b. Substance use disorder (except tobacco-related disorders/caffeine-related disorders) i. Alcohol consumption must be limited to ≤ 40 gram for men and ≤ 20 gram for women per day, e.g. ≤ two/one large beer (0.5 l) for men/women.
5. Use of classical psychedelics (i.e. LSD, psilocybin, mescaline, dimethyltryptamine) in the past year and or more than five life-time uses of classical psychedelics.
6. Failure to establish sufficient rapport with the two therapists as judged by them after the first two preparation sessions
7. Lithium intake
8. The patient has any disorder for which the treatment takes priority over treatment of depression or is likely to interfere with the study treatment or impair treatment compliance. This includes current signs/symptoms of liver or renal insufficiency, hypothyroidism or hyperthyroidism (subjects who are on stable treatment with thyroid supplementation and show an euthyroid metabolism with normal thyroid-stimulating hormone [TSH] may participate), significant cardiac disease (including current or past history of atrial fibrillation/flutter), vascular, pulmonary, endocrine, neurologic (including epilepsy), hematologic, inflammatory (e.g., rheumatoid arthritis, inflammatory bowel disease, Crohn's disease) or metabolic diseases as long as these diseases are not medically controlled or might significantly interfere with participation in the study. Diabetes mellitus (DM) may be allowed when blood glucose is stably controlled (HbA1c less than 7.5% or 58 mmol/mol).

   a. To rule out the presence of any serious neurological condition that might be underlying the depression (e.g. Parkinson's Disease, dementia), patients must provide a recent (i.e. not older than 5 years) brain neuroimaging (MRI or CT). If the clinical manifestation has changed qualitatively or in severity, a more recent neuroimaging is required.
9. Women who are pregnant, nursing or refuse to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) throughout their study participation. Women of childbearing potential must have a negative urine pregnancy test at screening and the two dosing days.
10. Positive urine drug screen for any illicit drugs of abuse or alcohol at any of the two dosing days. The regular drug screen includes cocaine, amphetamine, opiates, ecstasy, EDDP, cannabinoids, benzodiazepines and barbiturates.
11. The subject has a QTc interval > 450 ms (for men) or > 470 ms (for women) (Fridericia's correction) at screening or at baseline, as calculated by the ECG equipment and evaluated by the investigator.
12. The subject has received an investigational drug or used an invasive investigational medical device within 3 months before the first administration of the study drug or anticipates participation in another clinical trial until the primary endpoint.
13. The subject is unwilling or unable to undergo multiple venipunctures because of poor tolerability or lack of easy access.
14. The subject is unable to read and understand the patient information and the consent form, complete study-related procedures, and/or communicate with the study staff. Cognitive impairment that would render the informed consent invalid or limit the ability of the subject to comply with the study requirements also excludes from participation in the study.
15. The subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
16. Subject has had major surgery (e.g., requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study.
17. The subject has undergone electroconvulsive therapy (ECT) within twelve months prior to screening or treatment with ketamine or esketamine within six months prior to screening.
18. The subject has received any prior treatment with vagal nerve stimulation, or a deep brain stimulation device.
19. Subject is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Treatment Response (defined as a ≥ 50% drop in depressive symptom severity as measured by the Hamilton Rating Scale for Depression; HAM-D) | Baseline - 6 weeks after the first dose
  The HAM-D is a 21-item rating scale to assess the severity of depressive symptoms after a semi-structured clinical interview. Items are rated on a scale from 0 (absent) to 4. The total score is calculated by summing the first 17 items (HAM-D17) and ranges between 0 and 51.

SECONDARY OUTCOMES:
% change in HAM-D total score | Baseline - 1 day/1 week/6 weeks after the first dose
Treatment Response (defined as a ≥ 50% drop in depressive symptom severity as measured by the Hamilton Rating Scale for Depression; HAM-D) | Baseline - 1 day/1 week after the first dose
Treatment response (≥ 50% drop) and % change in HAM-D total score | Baseline - 12 weeks after the first dose
Treatment response (≥ 50% drop) and % change in the Beck Depression Inventory (BDI) - II | Baseline - 1 day/1 week/6 weeks after both doses
  The BDI is a reliable and valid 21-item self-rating questionnaire for the assessment of depressive symptoms. Patients rate their symptoms according to four severity ratings per item (0-3). The total score determines the severity of depression, differentiating between absent (0 - 9), mild (10 - 18), moderate (19 - 29) and severe (≥ 30) depression.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Gründer, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (2):
- Germany (2):
  - Charité Berlin, Campus Mitte, Department of Psychiatry and Psychotherapy, Berlin
  - Central Institute of Mental Health (CIMH), Mannheim

IPD SHARING:
Plan to Share IPD: Yes